CLINICAL TRIAL: NCT01207583
Title: Prevenar Post-Licensure Safety Study in Russia: Frequency Of Fever Post Vaccination
Brief Title: Prevenar (PCV-7) Post-Licensure Safety Study In Russia
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0887X1-4596; B1841011
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Children After Vaccination
Keywords: vaccine; infant; healthy subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy children after vaccination: healthy children after vaccination
  Interventions: Other: Non-interventional observational study

INTERVENTIONS:
Other: Non-interventional observational study — Non-interventional observational study

SUMMARY:
This study is planned to monitor the local and/or systemic reactions and compatibility of PCV-7 with routine vaccines in the Russian National immunization schedule. Consistent with the observational nature of this protocol, Prevenar will be administered as standard of care.

The aim of this study is to estimate the incidence of febrile reactions more than 38.0 degrees Celsius, specifically (≥38 to < 39 degrees C; > 39 to < 40 degrees C and > 40 degrees C, and the frequency of other local or systemic reactions following vaccination with Prevenar (PCV-7) co-administered with other routine childhood vaccines under the conditions of routine daily use in the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Infants eligible for Prevenar vaccination according to the Regulatory approved terms of the marketing authorization in the Russian Federation:
* Infants from 3 months up to 23 months of age who may benefit from active immunization against disease caused by Streptococcus pneumoniae serotypes 4, 6B, 9V, 14, 18C, 19F and 23F (including sepsis, meningitis, pneumonia, bacteraemia and acute otitis media).
* Parents or legal guardians willing and able to complete the diary cards.

Exclusion Criteria:

* Hypersensitivity to the active substances or to any of the excipients;
* Hypersensitivity to diphtheria toxoid;
* Age less than 3 months or greater than or equal to 2 years at enrollment;
* Contraindications as listed in the Package Insert / Russian SmPC for either Prevenar or for any concomitantly used other vaccines;
* Previously vaccinated with 23-valent pneumococcal polysaccharide vaccine;
* Prophylactic use of non-steroidal anti-inflammatory medications and/or acetaminophen (e.g., paracetamol). However, acetaminophen/paracetamol may be administered for treatment of fever, pain, etc.

Ages: 3 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants and Children from 3 months to 23 months at enrollment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Russia (4):
  - Russian State Medical University, Moscow
  - Russian Academy of Medical Sciences, Moscow
  - Research Institute of Childhood Infections, Saint Petersburg
  - City Children's Clinical Hospital #8, Yekaterinburg

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0887X1-4596&StudyName=Prevenar%20%28PCV-7%29%20Post-Licensure%20Safety%20Study%20In%20Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Cohort (3-6 Months): Participants in the age group 3-6 months received 4 doses (Dose 1, Dose 2, Dose 3 and Dose 4) of 7-valent pneumococcal conjugate vaccine (PCV7) as standard care as per the Summary of Product Characteristics (SmPC).
- Catch-up Cohort (7-11 Months): Participants in the age group 7-11 months received 3 doses (Dose 1, Dose 2 and Dose 3) of PCV7 vaccine as standard care as per the SmPC.
- Catch-up Cohort (12-23 Months): Participants in the age group 12-23 months received 2 doses (Dose 1 and Dose 2) of PCV7 vaccine as standard care as per the SmPC.
Period: Overall Study
Arm/Group | Primary Cohort (3-6 Months) | Catch-up Cohort (7-11 Months) | Catch-up Cohort (12-23 Months)
Started | 14 | 31 | 55
Dose 1 | 14 | 31 | 55
Dose 2 | 13 | 29 | 54
Dose 3 | 13 | 27 | 0
Dose 4 | 7 | 0 | 0
Completed | 13 | 26 | 54
Not Completed | 1 | 5 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Participant failed to return | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Primary Cohort (3-6 Months): Participants in the age group 3-6 months received 4 doses (Dose 1, Dose 2, Dose 3 and Dose 4) of PCV7 vaccine as standard care as per the SmPC.
- Total: Total of all reporting groups
Arm/Group | Primary Cohort (3-6 Months) | Catch-up Cohort (7-11 Months) | Catch-up Cohort (12-23 Months) | Total
Number analyzed (Participants) | 14 | 31 | 55 | 100
Age, Customized [Number; unit: Participants]
  3 to 6 months | 14 | 0 | 0 | 14
  7 to 11 months | 0 | 31 | 0 | 31
  12 to 23 months | 0 | 0 | 55 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 19 | 37
  Male | 9 | 18 | 36 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Febrile Reactions Post-dose 1
Description: Febrile reactions were defined as reactions which causes a rise in body temperature following vaccination in children. Fever was defined as a temperature of greater than or equal to (>=) 38 degrees Celsius (C). Percentage of participants with febrile reaction of >=38 degrees C to less than or equal to (<=) 39 degrees C, >39 degrees C to <=40 degrees C and >40 degrees C were observed.
Time Frame: Day 1 to Day 3 post-dose 1
Population: Safety set (post-dose 1) population included all participants who received Dose 1 and who had safety follow-up data following Dose 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Primary Cohort (3-6 Months): Participants in the age group 3-6 months received Dose 1 of PCV7 vaccine as standard care as per the SmPC.
- Catch-up Cohort (7-11 Months): Participants in the age group 7-11 months received Dose 1 of PCV7 vaccine as standard care as per the SmPC.
- Catch-up Cohort (12-23 Months): Participants in the age group 12-23 months received Dose 1 of PCV7 vaccine as standard care as per the SmPC.
Arm/Group | Primary Cohort (3-6 Months) | Catch-up Cohort (7-11 Months) | Catch-up Cohort (12-23 Months)
Number analyzed (Participants) | 14 | 31 | 55
Percentage of participants
  38 to 39 degrees C | 14.3 [4.0 to 39.9] | 16.1 [7.1 to 32.6] | 1.8 [0.3 to 9.6]
  >39 to 40 degrees C | 0.0 [0.0 to 21.5] | 3.2 [0.6 to 16.2] | 3.6 [1.0 to 12.3]

2. Primary Outcome: Percentage of Participants With Febrile Reactions Post-dose 2
Description: Febrile reactions were defined as reactions which causes a rise in body temperature following vaccination in children. Fever was defined as a temperature of >=38 degrees C. Percentage of participants with febrile reaction of >=38 degrees C to <=39 degrees C was observed.
Time Frame: Day 1 to Day 3 post-dose 2
Population: Safety set (post-dose 2) population included all participants who received Dose 2 and who had safety follow-up data following Dose 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Primary Cohort (3-6 Months): Participants in the age group 3-6 months received Dose 2 of PCV7 vaccine as standard care as per the SmPC.
- Catch-up Cohort (7-11 Months): Participants in the age group 7-11 months received Dose 2 of PCV7 vaccine as standard care as per the SmPC.
- Catch-up Cohort (12-23 Months): Participants in the age group 12-23 months received Dose 2 of PCV7 vaccine as standard care as per the SmPC.
Arm/Group | Primary Cohort (3-6 Months) | Catch-up Cohort (7-11 Months) | Catch-up Cohort (12-23 Months)
Number analyzed (Participants) | 13 | 29 | 54
Percentage of participants | 23.1 [8.2 to 50.3] | 10.3 [3.6 to 26.4] | 0.0 [0.0 to 6.6]

3. Primary Outcome: Percentage of Participants With Febrile Reactions Post-dose 3
Description: as for outcome 2
Time Frame: Day 1 to Day 3 post-dose 3
Population: Safety set (post-dose 3) population included all participants who received Dose 3 and who had safety follow-up data following Dose 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Primary Cohort (3-6 Months): Participants in the age group 3-6 months received Dose 3 of PCV7 vaccine as standard care as per the SmPC.
- Catch-up Cohort (7-11 Months): Participants in the age group 7-11 months received Dose 3 of PCV7 vaccine as standard care as per the SmPC.
Arm/Group | Primary Cohort (3-6 Months) | Catch-up Cohort (7-11 Months)
Number analyzed (Participants) | 13 | 26
Percentage of participants | 15.4 [4.3 to 42.2] | 0.0 [0.0 to 12.9]

4. Primary Outcome: Percentage of Participants With Febrile Reactions Post-dose 4
Description: Febrile reactions were defined as reactions which causes a rise in body temperature following vaccination in children. Fever was defined as a temperature of >=38 degrees C. Percentage of participants with febrile reaction of >=38 degrees C was observed.
Time Frame: Day 1 to Day 3 post-dose 4
Population: Safety set (post-dose 4) population included all participants who received Dose 4 and who had safety follow-up data following Dose 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Primary Cohort (3-6 Months): Participants in the age group 3-6 months received Dose 4 of PCV7 vaccine as standard care as per the SmPC.
Arm/Group | Primary Cohort (3-6 Months)
Number analyzed (Participants) | 7
Percentage of participants | 0.0 [0.0 to 35.4]

5. Secondary Outcome: Percentage of Participants With Pre-Specified Local Reactions Post-dose 1
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Induration and redness were scaled as Any (induration or redness present); Mild (<2.5 centimeters [cm]); Moderate (>=2.5 cm to <5.0 cm); Severe (>=5.0 cm). Participants may be represented in more than 1 category. Solicited local reactions included redness, swelling and tenderness while unsolicited local reactions included injection site hematoma, injection site hemorrhage, injection site induration and injection site warmth.
Time Frame: Day 1 to Day 3 post-dose 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Primary Cohort (3-6 Months) | Catch-up Cohort (7-11 Months) | Catch-up Cohort (12-23 Months)
Number analyzed (Participants) | 14 | 31 | 55
Percentage of participants
  Redness | 7.1 | 19.4 | 27.3
  Swelling | 0.0 | 6.5 | 25.5
  Tenderness | 7.1 | 29.0 | 23.6
  Injection site hematoma | 0.0 | 0.0 | 1.8
  Injection site hemorrhage | 0.0 | 3.2 | 1.8
  Injection site induration | 7.1 | 0.0 | 0.0
  Injection site warmth | 0.0 | 0.0 | 1.8

6. Secondary Outcome: Percentage of Participants With Pre-Specified Local Reactions Post-dose 2
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Induration and redness were scaled as Any (induration or redness present); Mild (<2.5 cm); Moderate (>=2.5 cm to <5.0 cm); Severe (>=5.0 cm). Participants may be represented in more than 1 category. Solicited local reactions included redness, swelling and tenderness while unsolicited local reactions included injection site hematoma, injection site hemorrhage, injection site induration and injection site warmth.
Time Frame: Day 1 to Day 3 post-dose 2
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Primary Cohort (3-6 Months) | Catch-up Cohort (7-11 Months) | Catch-up Cohort (12-23 Months)
Number analyzed (Participants) | 13 | 29 | 54
Percentage of participants
  Redness | 23.1 | 13.8 | 20.4
  Swelling | 0.0 | 0.0 | 11.1
  Tenderness | 0.0 | 6.9 | 16.7
  Injection site hemorrhage | 0.0 | 0.0 | 3.7
  Injection site induration | 0.0 | 0.0 | 1.9

7. Secondary Outcome: Percentage of Participants With Pre-Specified Local Reactions Post-dose 3
Description: as for outcome 6
Time Frame: Day 1 to Day 3 post-dose 3
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Primary Cohort (3-6 Months) | Catch-up Cohort (7-11 Months)
Number analyzed (Participants) | 13 | 26
Percentage of participants
  Redness | 15.4 | 3.8
  Swelling | 7.7 | 3.8
  Tenderness | 7.7 | 7.7
  Injection site induration | 7.7 | 0.0

8. Secondary Outcome: Percentage of Participants With Pre-Specified Local Reactions Post-dose 4
Description: as for outcome 6
Time Frame: Day 1 to Day 3 post-dose 4
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Primary Cohort (3-6 Months)
Number analyzed (Participants) | 7
Percentage of participants
  Redness | 14.3
  Swelling | 14.3
  Injection site induration | 14.3

9. Secondary Outcome: Percentage of Participants With Pre-Specified Systemic Events Post-dose 1
Description: Systemic events (any fever >=38 degrees C, decreased appetite, diarrhea, restless sleep, unusual crying, unusual fussiness, unusual irritability, and vomiting) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Day 1 to Day 3 post-dose 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Catch-up Cohort (12-23 Months): Participants in the age group 12-23 months received Dose 1 of PCV7 vaccines as standard care as per the SmPC.
Arm/Group | Primary Cohort (3-6 Months) | Catch-up Cohort (7-11 Months) | Catch-up Cohort (12-23 Months)
Number analyzed (Participants) | 14 | 31 | 55
Percentage of participants
  Decreased appetite | 7.1 | 19.4 | 23.6
  Diarrhea | 7.1 | 3.2 | 9.1
  Fever | 14.3 | 19.4 | 5.5
  Restless sleep | 7.1 | 32.3 | 27.3
  Unusual crying | 14.3 | 25.8 | 30.9
  Unusual fussiness | 7.1 | 6.5 | 12.7
  Unusual irritability | 21.4 | 19.4 | 25.5
  Vomiting | 0.0 | 6.5 | 3.6

10. Secondary Outcome: Percentage of Participants With Pre-Specified Systemic Events Post-dose 2
Description: as for outcome 9
Time Frame: Day 1 to Day 3 post-dose 2
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Primary Cohort (3-6 Months) | Catch-up Cohort (7-11 Months) | Catch-up Cohort (12-23 Months)
Number analyzed (Participants) | 13 | 29 | 54
Percentage of participants
  Decreased appetite | 15.4 | 10.3 | 9.3
  Diarrhea | 15.4 | 3.4 | 0.0
  Fever | 23.1 | 10.3 | 0.0
  Restless sleep | 23.1 | 24.1 | 16.7
  Unusual crying | 23.1 | 20.7 | 13.0
  Unusual fussiness | 15.4 | 6.9 | 7.4
  Unusual irritability | 23.1 | 6.9 | 9.3
  Vomiting | 7.7 | 0.0 | 1.9

11. Secondary Outcome: Percentage of Participants With Pre-Specified Systemic Events Post-dose 3
Description: as for outcome 9
Time Frame: Day 1 to Day 3 post-dose 3
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Primary Cohort (3-6 Months) | Catch-up Cohort (7-11 Months)
Number analyzed (Participants) | 13 | 26
Percentage of participants
  Decreased appetite | 7.7 | 0.0
  Diarrhea | 15.4 | 3.8
  Fever | 15.4 | 0.0
  Restless sleep | 46.2 | 11.5
  Unusual crying | 15.4 | 11.5
  Unusual fussiness | 15.4 | 0.0
  Unusual irritability | 7.7 | 7.7
  Vomiting | 15.4 | 3.8

12. Secondary Outcome: Percentage of Participants With Pre-Specified Systemic Events Post-dose 4
Description: as for outcome 9
Time Frame: Day 1 to Day 3 post-dose 4
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Primary Cohort (3-6 Months)
Number analyzed (Participants) | 7
Percentage of participants
  Restless sleep | 28.6
  Unusual crying | 14.3
  Unusual irritability | 14.3

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Dose 1 (Primary Cohort [3-6 Months]): Participants in the age group 3-6 months received Dose 1 of PCV7 vaccine as standard care as per the SmPC.
- Dose 2 (Primary Cohort [3-6 Months]): Participants in the age group 3-6 months received Dose 2 of PCV7 vaccine as standard care as per the SmPC.
- Dose 3 (Primary Cohort [3-6 Months]): Participants in the age group 3-6 months received Dose 3 of PCV7 vaccine as standard care as per the SmPC.
- Dose 4 (Primary Cohort [3-6 Months]): Participants in the age group 3-6 months received Dose 4 of PCV7 vaccine as standard care as per the SmPC.
- Dose 1 (Catch-up Cohort [7-11 Months]): Participants in the age group 7-11 months received Dose 1 of PCV7 vaccine as standard care as per the SmPC.
- Dose 2 (Catch-up Cohort [7-11 Months]): Participants in the age group 7-11 months received Dose 2 of PCV7 vaccine as standard care as per the SmPC.
- Dose 3 (Catch-up Cohort [7-11 Months]): Participants in the age group 7-11 months received Dose 3 of PCV7 vaccine as standard care as per the SmPC.
- Dose 1 (Catch-up Cohort [12-23 Months]): Participants in the age group 12-23 months received Dose 1 of PCV7 vaccine as standard care as per the SmPC.
- Dose 2 (Catch-up Cohort [12-23 Months]): Participants in the age group 12-23 months received Dose 2 of PCV7 vaccine as standard care as per the SmPC.
Arm/Group | Dose 1 (Primary Cohort [3-6 Months]) | Dose 2 (Primary Cohort [3-6 Months]) | Dose 3 (Primary Cohort [3-6 Months]) | Dose 4 (Primary Cohort [3-6 Months]) | Dose 1 (Catch-up Cohort [7-11 Months]) | Dose 2 (Catch-up Cohort [7-11 Months]) | Dose 3 (Catch-up Cohort [7-11 Months]) | Dose 1 (Catch-up Cohort [12-23 Months]) | Dose 2 (Catch-up Cohort [12-23 Months])
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13 | 0/7 | 1/31 | 0/29 | 0/26 | 1/55 | 0/54
Other Adverse Events (participants affected / at risk) | 6/14 | 6/13 | 6/13 | 2/7 | 17/31 | 8/29 | 5/26 | 27/55 | 16/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose 1 (Primary Cohort [3-6 Months]) (N=14) | Dose 2 (Primary Cohort [3-6 Months]) (N=13) | Dose 3 (Primary Cohort [3-6 Months]) (N=13) | Dose 4 (Primary Cohort [3-6 Months]) (N=7) | Dose 1 (Catch-up Cohort [7-11 Months]) (N=31) | Dose 2 (Catch-up Cohort [7-11 Months]) (N=29) | Dose 3 (Catch-up Cohort [7-11 Months]) (N=26) | Dose 1 (Catch-up Cohort [12-23 Months]) (N=55) | Dose 2 (Catch-up Cohort [12-23 Months]) (N=54)
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose 1 (Primary Cohort [3-6 Months]) (N=14) | Dose 2 (Primary Cohort [3-6 Months]) (N=13) | Dose 3 (Primary Cohort [3-6 Months]) (N=13) | Dose 4 (Primary Cohort [3-6 Months]) (N=7) | Dose 1 (Catch-up Cohort [7-11 Months]) (N=31) | Dose 2 (Catch-up Cohort [7-11 Months]) (N=29) | Dose 3 (Catch-up Cohort [7-11 Months]) (N=26) | Dose 1 (Catch-up Cohort [12-23 Months]) (N=55) | Dose 2 (Catch-up Cohort [12-23 Months]) (N=54)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disbacteriosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 3
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Crying (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Redness (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 1 | 6 | 4 | 1 | 15 | 11
Swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 14 | 6
Tenderness (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 9 | 2 | 2 | 13 | 9
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Injection site induration (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Injection site warmth (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (General disorders) | 1 | 2 | 1 | 0 | 6 | 3 | 0 | 13 | 5
Diarrhea (General disorders) | 1 | 2 | 2 | 0 | 1 | 1 | 1 | 5 | 0
Fever (General disorders) | 2 | 3 | 2 | 0 | 6 | 3 | 0 | 3 | 0
Restless sleep (General disorders) | 1 | 3 | 6 | 2 | 10 | 7 | 3 | 15 | 9
Unusual crying (General disorders) | 2 | 3 | 2 | 1 | 8 | 6 | 3 | 17 | 7
Unusual fussiness (General disorders) | 1 | 2 | 2 | 0 | 2 | 2 | 0 | 7 | 4
Unusual irritability (General disorders) | 3 | 3 | 1 | 1 | 6 | 2 | 2 | 14 | 5
Vomiting (General disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.